CLINICAL TRIAL: NCT00807872
Title: Radioimmunoimaging (PET/CT) of Patients With AL Amyloidosis Using the 124I-Labeled Amyloid-Reactive Monoclonal Antibody Mu 11-1F4
Brief Title: Radioimmunoimaging of AL Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alan Solomon, Alan Solomon, M.D., University of Tennessee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2625; NCT00808847 (obsolete NCT alias)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Primary Amyloidosis
Keywords: Radioimmunoimaging; AL Amyloidosis; PET/CT
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I-124 Mu 11-1F4 sterile injection (Other): Single arm study
  Interventions: Biological: 124I-labeled monoclonal antibody Mu 11-1F4

INTERVENTIONS:
Biological: 124I-labeled monoclonal antibody Mu 11-1F4 — Single infusion of radiolabeled antibody: 2 mCi (1 mg)
  Other Names: anti-amyloid radioimmunoimaging agent

SUMMARY:
The purpose of the study is to determine the capability of a radiolabeled amyloid-reactive monoclonal antibody to document the presence and distribution of amyloid deposits by PET/CT imaging in patients with AL amyloidosis.

DETAILED DESCRIPTION:
To be eligible for this study, patients must have a confirmed diagnosis of AL amyloidosis without significant cardiac (New York Heart Association class IV) disease and not be on kidney dialysis. Additionally, after testing, their blood must not contain antibodies to mouse proteins. The study requires an intravenous infusion, given over 10 minutes, of the radiolabeled antibody, followed 48 hours later by a PET/CT scan. A repeat scan is done 5 to 7 days after infusion of the antibody. A 5 ml blood specimen needs to be furnished 4 and 8 weeks after the antibody infusion.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AL amyloidosis

Exclusion Criteria:

* New York Heart Association class IV
* patient on renal dialysis
* serum antibodies to mouse protein

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Radioimmunoimaging of AL amyloid deposits by PET/CT | 10-14 days post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Alan Solomon, MD, Principal Investigator — University of Tennessee Graduate School of Medicine
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

REFERENCES:
- [Derived] Wall JS, Kennel SJ, Stuckey AC, Long MJ, Townsend DW, Smith GT, Wells KJ, Fu Y, Stabin MG, Weiss DT, Solomon A. Radioimmunodetection of amyloid deposits in patients with AL amyloidosis. Blood. 2010 Sep 30;116(13):2241-4. doi: 10.1182/blood-2010-03-273797. Epub 2010 Jun 3. PMID 20522711
- See also: Amyloid Research Foundation — http://www.amyloidosisresearchfoundation.org/